CLINICAL TRIAL: NCT00006175
Title: Cytokine Responses to Acute Inflammation in the Oral Surgery Model
Brief Title: Cyclooxygenase Levels Following Surgery to Remove Third Molars (Wisdom Teeth)
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000190; 00-D-0190
Record Dates: First submitted 2000-08-12; First posted 2000-08-14 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-10

CONDITIONS: Healthy; Inflammation
Keywords: Cyclooxygenase; COX-1; COX-2; Prostanoids; P.C.R.; Healthy Volunteer
MeSH Terms: conditions — Inflammation

SUMMARY:
This study will measure levels of an enzyme called cyclooxygenase in gum tissue following third molar (wisdom tooth) extraction. Cyclooxygenase is thought to contribute to pain that normally follows tissue injury or surgery.

Healthy volunteers between 16 and 35 years of age who require removal of their third molars may be eligible for this study. Participants will receive an injection of a local anesthetic (lidocaine) in the mouth and a sedative (midazolam) through an arm vein before surgery. Before the tooth is removed, a small tissue sample (biopsy) will be collected from the gum tissue covering one of the lower third molars to be extracted. After surgery, a second biopsy will be taken at some point between just after surgery to the time when pain from the extraction starts to develop. These tissue samples will be analyzed for cyclooxygenase levels.

Patients will stay in the clinic for up to 4 hours after surgery while the anesthetic wears off. During this time, they will complete pain questionnaires. If needed, patients may receive additional medicine for pain relief at any time during the surgery or the 4-hour observation period. They will also be given standard pain medication to take home at the end of the study.

DETAILED DESCRIPTION:
Prostanoids are inflammatory mediators that have been implicated in all stages of acute and chronic inflammation. The inhibition of prostanoid synthesis by NSAIDs forms the basis of their therapeutic as well as side effects. NSAIDs directly inhibit cyclooxygenase [COX], which leads to reduction of prostaglandin synthesis but also to gastric erosions, inhibition of platelet aggregation and nephrotoxicity. The identification of the two isoforms of COX lead to the hypothesis that COX-2 is responsible for the production of prostaglandins following tissue injury, while COX-1 is involved in normal homeostasis. This hypothesis is primarily based on the results of animal studies and chronic inflammatory conditions such as arthritis. Recent results in the oral surgery model of acute inflammation suggest that COX-2 is present in the oral mucosa and may contribute to prostanoid production during acute inflammation rather than require induction in response to the injury. The proposed study aims to evaluate the time course of COX-1 and COX-2 in acute inflammation by evaluating levels of mRNA at baseline prior to surgery, at the completion of surgery, and at one, two and three hours following surgery.

ELIGIBILITY:
INCLUSION CRITERIA:

Subjects will be healthy volunteers between the ages 16-35 years presenting to the Clinical Center for removal of their third molars.

The type of third molar will be characterized at the time of screening by oral exam and panoramic radiograph:

1. Erupted tooth: Clinical crown is present in the mouth and is not covered by soft tissue.
2. Soft tissue impaction: Clinical crown is not present in the mouth but the adjacent alveolar bone does not cover any portion of the crown in the radiograph.
3. Partial bony impaction: Clinical crown is not present in the mouth and the alveolar bone covers some but not all of the crown in the radiograph.
4. Full bony impaction: Clinical crown is not present in the mouth and the alveolar bone covers most or all of the crown in the radiograph.

Patients will be eligible for inclusion in this study if the two mandibular molars are classified as partial or full bony impactions.

EXCLUSION CRITERIA:

Patients who are pregnant or nursing.

Presence of infection or inflammation [pericoronitis] at either extraction site.

Patients who are taking any of the following drugs: anti-depressants, diuretics, aspirin on a near daily basis, coumadin or other blood thinners; or other drugs that might influence pain report or COX formation, e.g. steroids.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160
Dates: Start 2000-08; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Smith CJ, Zhang Y, Koboldt CM, Muhammad J, Zweifel BS, Shaffer A, Talley JJ, Masferrer JL, Seibert K, Isakson PC. Pharmacological analysis of cyclooxygenase-1 in inflammation. Proc Natl Acad Sci U S A. 1998 Oct 27;95(22):13313-8. doi: 10.1073/pnas.95.22.13313. PMID 9789085
- [Background] Pairet M, van Ryn J. Experimental models used to investigate the differential inhibition of cyclooxygenase-1 and cyclooxygenase-2 by non-steroidal anti-inflammatory drugs. Inflamm Res. 1998 Oct;47 Suppl 2:S93-101. doi: 10.1007/s000110050289. PMID 9831330
- [Background] Morrison BW, Christensen S, Yuan W, Brown J, Amlani S, Seidenberg B. Analgesic efficacy of the cyclooxygenase-2-specific inhibitor rofecoxib in post-dental surgery pain: a randomized, controlled trial. Clin Ther. 1999 Jun;21(6):943-53. doi: 10.1016/S0149-2918(99)80016-2. PMID 10440619